CLINICAL TRIAL: NCT00348413
Title: Comparison of Efficacy and Safety of Intravenous Pulsed Methylprednisolone and Oral Methotrexate Versus Intravenous Pulsed Methylprednisolone and Oral Placebo in the Treatment of Active Moderate and Severe Thyroid Eye Disease - a Prospective, Randomized, Double-blind, Parallel, Controlled Multidisciplinary Clinical Trial and Imaging Study.
Brief Title: Thyroid Treatment Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: International Stem Cell Forum (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R272/16/2002
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves ophthalmopathy/therapy; Randomized controlled trial; Methylprednisolone; Methotrexate
MeSH Terms: conditions — Graves Ophthalmopathy

INTERVENTIONS:
Drug: Intravenous Methylprednisolone + Oral Methotrexate vs Intravenous Methylprednisolone + Placebo

SUMMARY:
This project will compare the efficacy and safety of 2 methods of disease modification in the treatment of active moderate and severe thyroid orbitopathy. A prospective, randomized, double-blind, parallel, controlled multidisciplinary clinical trial involving Singapore National Eye Centre, National University Hospital, Changi General Hospital, Tan Tock Seng Hospital and University of British Columbia Orbital Services, Singapore Eye Research Institute, Singapore General Hospital Endocrinology and Radiology Departments and Tan Tock Seng Hospital Rheumatology Department is planned. The SingHealth-SGH High Field MR Research Laboratory will be involved in the MR imaging of the trial patients.

Patients who satisfy the inclusion and exclusion criteria will be asked to participate in this trial. After informed consent (Appendix B) is obtained, each patient will be randomized into one of two treatment arms: 1) Intravenous high-dose pulsed methylprednisolone (1 gram infusion over 1 hour per day with a total of 3 doses over 3 days; 4 cycles at 6 weekly intervals) and oral placebo and 2) Intravenous high-dose pulsed methylprednisolone (same dose) plus oral methotrexate 7.5 mg per week for 2 weeks, increased to 10 mg per week for another 2 weeks then 12.5 mg per week for 5 months (total 6 months of methotrexate treatment). Depending on patient response, the dose can be further increased by 2.5mg per week every 4 weeks to a maximum of 20 mg per week. A strict management protocol will be observed for each recruited patient. Patients who develop adverse side effects or need for surgical intervention will receive appropriate treatment (i.e. treatment will deviate from the protocol but will continue to be monitored). Patients who refuse treatment will be observed clinically and with imaging as a natural control group until such time as intervention is accepted.

The patients will have a baseline assessment followed by regular visits to assess treatment response and adverse effects. Observations will include the use of an inflammatory index, motility measurements including quantitative ductions, exophthalmometry readings, palpebral aperture readings and indices of optic nerve function. With regards to the imaging, the patients will be assessed with an initial quantitative CT scan and 3-Tesla MRI scan prior to treatment. After treatment is started, patients will also undergo repeat MRI scan at 24 weeks and 72 weeks to assess quantitative changes with treatment using the Muscle Diameter Index (MDI) and Pixel Value Ratio (PVR) for the inferior rectus, superior rectus, the medial rectus, lateral rectus and orbital fat (Appendix E). Serum and urine will be obtained at the same time intervals as the MRI scan to assess levels of thyroid hormones, thyroid antibodies and urinary glycosaminoglycans (GAGs). Free T4, free T3 and TSH will be recorded to monitor control of hyperthyroidism. Thyroid antibodies measured will include thyroid stimulating immunoglobulin (TSI), thyrotropin-binding inhibition antibody (TB II), thyroid peroxidase antibodies and thyroglobulin antibody. Other tests including the full blood count, urea and electrolytes will be run prior to each dose of steroid treatment and during follow-up to monitor for adverse effects.

The results of the assessments will be analyzed for significant differences in treatment response between the 2 groups. The indices of interest will include the percentage of patients in each group who demonstrate a decrease in the inflammatory index of at least 2 points and the time taken for 50% of patients to show such a decrease. Other parameters that reflect the visual function and motility will be compared at different points in time after starting treatment to observe response and sustainability of response. From the serial MRI scans, quantitative analysis of orbital tissues will be done to identify changes with treatment. Antibody and GAG levels will be analyzed to detect any change with treatment. The types and frequency of adverse side effects in the 2 groups will also be assessed.

80 normal subjects will be recruited for MRI scan of the orbits and brain to obtain normative values for the MDI and PVR for the Asian population (Appendix E). This will include 20 subjects from each of 4 decades (21-30 years, 31-40 years, 41-50 years, 51-60 years).

The normative data will also be used to create a virtual orbital atlas. This aspect of the study will be performed in collaboration with the Labs for Information Technology (A-Star).

DETAILED DESCRIPTION:
Since 1835 when Graves first described the eye changes in thyroid disease, considerable literature on investigating the basic disease process, the clinical behaviour, natural history and various medical and surgical treatments on thyroid orbitopathy has developed.

3.1 Pathogenesis 11, 12

HLA-DR histocompatibility loci which play a role in T-cell response have been associated with thyroid orbitopathy but no specific gene has been identified as yet.

It is believed that TSH receptors may be the autoantigen in Graves' hyperthyroidism, orbitopathy and pretibial myxoedema. Somehow, T-lymphocytes are activated and proceed to infiltrate orbital and other soft tissues. This sets off cytokine release which together with oxygen free radicals and fibrogenic growth factors leads to increased hydrophilic glycosaminoglycan (GAG) synthesis and pre-adipocyte transformation. The overall effect is an increase in orbital muscle and fat volume and inflammatory oedema which ultimately may result in muscle fibrosis and optic nerve compression.

3.2 Pathology

The histopathological features correlate with the immunogenetic theory in thyroid orbitopathy. The extraocular muscles are infiltrated by lymphocytes, macrophages, plasma cells and mast cells. Hydrophilic mucopolysaccharides are deposited and are seen separating the muscle bundles and fibres. In the later stages, fibrosis and muscle degeneration with fat replacement is noted.

3.3 Clinical Features

Based on literature review and the experience of the University of Columbia Orbital Clinic which saw over 2000 cases from 1976 to 2002.

1. Indices of disease activity (largely subjective)

   * Acuity of onset and progression

     * Acute (within a week) or subacute (3 months or under 3 months) or chronic onset (over 3 months)
     * Slow or rapid development (progression)
   * Subjective symptoms

     * Spontaneous retrobulbar pain
     * Pain on extraocular movement
   * Soft tissue features

     - Swelling, injection and chemosis noted by the patient
   * Patient assessment of symptoms and signs - Same, better or worse
2. Indices of disease severity and extent (largely objective)

   * Lid and conjunctival swelling
   * Extraocular muscle function
   * Proptosis
   * Optic nerve function
   * Imaging changes in orbital tissues The NOSPECS classification of thyroid orbitopathy 13,14 does not give a clear picture of disease activity and severity. It does not guide prognostication and management and is thus abandoned in favour of the above assessment which looks specifically at indices which allow one to judge whether the disease is active and how severe it is 1.

From such an assessment, a treatment algorithm can be formulated:

3.4 Current Treatment

Although the exact aetiology and pathophysiology of thyroid orbitopathy remains unclear, what is known about the disease suggests an autoimmune mechanism at work 1,2. The initial phase of the disease is marked by clinical inflammatory changes and is followed by quiescence during which cicatricial and persistent orbital volume changes are more pronounced. In this latter phase, surgery alone works to alleviate symptoms. To avoid these end-stage developments, the disease should be treated during the active stage.

A recent trend in the management of thyroid orbitopathy has been to treat active disease with intravenous pulsed methylprednisolone 1,3-8. This step away from oral steroids arose from a desire to avoid the many known complications of prolonged oral steroid use as well as perceived lower success rates with the use of oral steroids. Marcocci et al 9 published in August 2001 results of a prospective, single-blind, randomized study that compared the effectiveness and tolerability of intravenous or oral glucocorticoids in association with orbital radiotherapy in the treatment of severe Graves' ophthalmopathy. This and other studies found that both treatments were effective (60-85% showing improvement) with the intravenous route associated with a lower rate of side effects. 3,4,5,6,7,9 Another treatment was reported by Smith and Rosenbaum in the British Journal of Ophthalmology 10. They described the use of oral methotrexate in the management of non-infectious orbital inflammatory disease. In their study, there were 3 patients with recalcitrant thyroid orbitopathy who had previously been treated with oral prednisolone, irradiation and surgical decompression. Two were still on oral prednisolone when oral methotrexate was started. All 3 showed clinical benefit and the 2 who were also on steroids initially were eventually able to cease steroid use. The good response may well be due to the fact that methotrexate, with its T-cell inhibiting effect, succeeded in halting the disease process especially when used together with corticosteroid.

The current treatment for those with progressively worse moderate or severe disease is medical decompression with either corticosteroid with or without cyclosporin or immunosuppressive agents such as methotrexate, cyclophosphamide or azathioprine as adjuvant therapy. The use of these latter agents are not well studied. When the soft tissue inflammation and orbital congestion is relieved, surgical redress of mechanical problems follows.

The role of radiotherapy remains unclear 15. Gorman et al conducted a prospective, randomized double-blind, placebo-controlled study of orbital radiotherapy for Graves' ophthalmopathy which failed to demonstrate any beneficial therapeutic effect 16. However, the study was flawed by the broad patient inclusion criteria and initiation of radiotherapy at different stages of the disease. Other studies have reported effective use of radiotherapy in the treatment of Graves' ophthalmopathy. Mourits conducted a randomized placebo-controlled trial which showed that external beam irradiation produced improvement in ocular motility in patients with mild or moderate disease 17.

We propose that active moderate and severe thyroid orbitopathy can be treated more aggressively with intravenous pulsed methylprednisolone and oral methotrexate in order to better stabilise the disease process and prevent cicatricial or compressive events. The question that this study aims to answer is whether this is a better treatment option compared to the current treatment in terms of efficacy and safety. Assessing the antibody and urinary GAG levels will yield information on serum and urinary profiles during treatment. We previously reported associations between thyroid autoantibodies and ophthalmopathy 18. The study will also use a 3-Tesla MRI to obtain normative values (MDI and PVR) for the Asian population and to evaluate quantitative changes in thyroid-related orbitopathy. This will provide a framework to study other multimodality therapy, including T-cell suppression, specific immunoglobulins and antifibroblastic agents.

4. STUDY PURPOSE

The purpose of this study is to investigate the effectiveness and safety of combined intravenous steroid and oral methotrexate in the treatment of patients with active moderate or severe thyroid orbitopathy. A prospective, randomized, double-blind, parallel, controlled clinical trial designed with this aim will provide useful information to aid future multimodality trials. This concept is based on the trend in managing rheumatologic disorders where early aggressive targeted multimodality therapy has improved treatment. The results of this study will also complement a planned radiotherapy study at the University of British Columbia

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed TED (as defined by Bartley and Gorman19)

   - Eyelid retraction (upper eyelid margin at or above the superior corneoscleral limbus in primary gaze without frontalis muscle contraction) in association with any one of the following:
   * Thyroid dysfunction or abnormal regulation (increased serum thyroxine or triiodothyronine level, decreased serum thyroid stimulating hormone level, absence of thyroid radioiodine uptake suppression after administration of triiodothyronine, or the presence of thyroid stimulating immunoglobulins in serum)
   * Exophthalmos (Hertel measurement of at least 20mm)
   * Extraocular muscle involvement (restrictive myopathy or objective evidence of enlarged muscles)
   * Optic nerve dysfunction (abnormal visual acuity, colour vision, pupillary reaction or perimetry not attributable to other causes)

   OR

   - Thyroid dysfunction or abnormal regulation in association with any one of the following:

   -Exophthalmos

   - Extraocular muscle involvement

   - Optic nerve dysfunction
2. Active disease

Inflammatory Index

Inflammatory Index

Soft tissue feature Rating Chemosis 0 Absent

1. Moderate (up to lid margin)
2. Severe (over lid margin; persists on closing eye)

Conjunctival injection 0 Absent 1 Present

Lid injection 0 Absent

1 Present

Lid edema 0 Absent

1. Moderate
2. Severe (festoons, overhang)

Pain at rest (clearly defined as retrobulbar aching) 0 Absent 1 Present

Pain on movement 0 Absent

1 Present

Total possible 8

Active disease is defined as an inflammatory index of at least 3 together with acute or subacute onset (3 months and under) and/or evidence of progression (from history or clinical observation).

(3) Moderate or severe disease

Primary Criteria

Mild Moderate Severe Inflammatory Index <3 3-5 >5

Motility <1/3 1/3 to 2/3 >2/3 (involving any one muscle) limitation limitation Limitation

Elevation, depression, adduction and abduction of the individual eyes will be measured with a modified Aimarck perimeter with input from both patient and the orthoptist who performs the test 20.

Secondary Criteria 21,22,23,24

Mild Moderate Severe Exophthalmos (mm) <21 21-24 25 or more

Best corrected vision (Logmar) - - 0.6 or worse

CT criterion (Muscle Diameter Index) 21-24 25-30 31 and above

These criteria are not considered absolutes and emphasize measurable indices based on previous studies.

The presence of at least 1 primary criterion and at least 1 secondary criterion places the patient in the more advanced disease group (in the situation where 1 primary criterion is mild and the other severe, the presence of 1 severe secondary criterion will yield a severe grade whereas absence of this criterion will result in a mild grade) eg 1) a patient with an inflammatory index of 6 and moderate limitation of extraocular motility, 21mm proptosis, 0.3 vision and MDI of 26 has moderate disease as the secondary criteria for severe disease was not present eg 2) a patient with an inflammatory index of 5 and mild limitation of extraocular motility, 21mm proptosis, 0.3 vision and MDI of 30 has moderate disease as 1 primary and 2 secondary criteria for moderate disease were present eg 3) a patient with inflammatory index of 6 and mild limitation of extraocular motility, 20mm proptosis, 0.3 vision and MDI of 21 has mild disease as the secondary criterion for severe disease was absent and the other primary parameter (motility) was graded mild.

(4) Age between 21 - 60

(5) Written informed consent is obtained

Exclusion Criteria:

1. Previous treatment for TED

   * Oral steroids (e.g. immunosuppressive dose) for last 3 months, radiotherapy
   * Intravenous pulsed steroid or methrotrexate therapy
2. Medically unfit to receive I/V high-dose pulsed methylprednisolone or methotrexate

   * History of cardiac arrthymias, recent acute myocardial infarction
   * History of seizure
   * History of acute bleeding peptic ulcer
   * History of pulmonary tuberculosis, Hepatitis B carrier, Hepatitis C positivity, HIV
   * Uncontrolled diabetes or hypertension (to be eligible for the trial, random blood glucose must be < 11.1 mmol/L and blood pressure must be 140/90 or lower#. If above these limits, patients can be treated and reviewed at 2 weeks for enrolment when criteria are met - provided the patient does not have optic neuropathy)
   * Hepatic dysfunction (Alb, AST, ALT and Alkaline phosphates levels must be within normal range for eligibility)
   * Renal impairment (Urea and Creatinine levels must be within normal range)
   * Abnormal blood count (outside normal range)
3. Others

   * Fertile females considering becoming pregnant during the course of the study and those not willing to take precautions to avoid pregnancy
   * Both female and male planning to start a family during the trial period or within 6 months of stopping the drugs
   * History of seizure
   * History of mental / psychiatric disorder
   * Patients with clinical features of optic nerve disc pallor at primary presentation will be excluded

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Inflammatory index

SECONDARY OUTCOMES:
Motility
Proptosis

CONTACTS AND LOCATIONS:
Overall Officials: Lay Leng Seah, MMed(Ophth), FRCS(Ed), Study Chair — Singapore National Eye Centre; Audrey Lee Geok Looi, MMed(Ophth), FRCS(Ed), Principal Investigator — Singapore National Eye Centre; Jack Rootman, MD. FRCS(C), Principal Investigator — University of British Columbia
Locations (1):
- Singapore National Centre, Singapore, Singapore

REFERENCES:
- [Background] Warwar RE. New insights into pathogenesis and potential therapeutic options for Graves orbitopathy. Curr Opin Ophthalmol. 1999 Oct;10(5):358-61. doi: 10.1097/00055735-199910000-00014. PMID 10621552
- [Background] Nagayama Y, Izumi M, Kiriyama T, Yokoyama N, Morita S, Kakezono F, Ohtakara S, Morimoto I, Okamoto S, Nagataki S. Treatment of Graves' ophthalmopathy with high-dose intravenous methylprednisolone pulse therapy. Acta Endocrinol (Copenh). 1987 Dec;116(4):513-8. doi: 10.1530/acta.0.1160513. PMID 3321820
- [Background] Kendall-Taylor P, Crombie AL, Stephenson AM, Hardwick M, Hall K. Intravenous methylprednisolone in the treatment of Graves' ophthalmopathy. BMJ. 1988 Dec 17;297(6663):1574-8. doi: 10.1136/bmj.297.6663.1574. PMID 2906260
- [Background] Guy JR, Fagien S, Donovan JP, Rubin ML. Methylprednisolone pulse therapy in severe dysthyroid optic neuropathy. Ophthalmology. 1989 Jul;96(7):1048-52; discussion 1052-3. doi: 10.1016/s0161-6420(89)32784-9. PMID 2771352
- [Background] Hiromatsu Y, Tanaka K, Sato M, Kuroki T, Nonaka K, Kojima K, Nishimura H, Nishida H, Kaise N. Intravenous methylprednisolone pulse therapy for Graves' ophthalmopathy. Endocr J. 1993 Feb;40(1):63-72. doi: 10.1507/endocrj.40.63. PMID 7951498
- [Background] Koshiyama H, Koh T, Fujiwara K, Hayakawa K, Shimbo S, Misaki T. Therapy of Graves' ophthalmopathy with intravenous high-dose steroid followed by orbital irradiation. Thyroid. 1994 Winter;4(4):409-13. doi: 10.1089/thy.1994.4.409. PMID 7711503
- [Background] Tagami T, Tanaka K, Sugawa H, Nakamura H, Miyoshi Y, Mori T, Nakao K. High-dose intravenous steroid pulse therapy in thyroid-associated ophthalmopathy. Endocr J. 1996 Dec;43(6):689-99. doi: 10.1507/endocrj.43.689. PMID 9075609
- [Background] Marcocci C, Bartalena L, Tanda ML, Manetti L, Dell'Unto E, Rocchi R, Barbesino G, Mazzi B, Bartolomei MP, Lepri P, Cartei F, Nardi M, Pinchera A. Comparison of the effectiveness and tolerability of intravenous or oral glucocorticoids associated with orbital radiotherapy in the management of severe Graves' ophthalmopathy: results of a prospective, single-blind, randomized study. J Clin Endocrinol Metab. 2001 Aug;86(8):3562-7. doi: 10.1210/jcem.86.8.7737. PMID 11502779
- [Background] Smith JR, Rosenbaum JT. A role for methotrexate in the management of non-infectious orbital inflammatory disease. Br J Ophthalmol. 2001 Oct;85(10):1220-4. doi: 10.1136/bjo.85.10.1220. PMID 11567968
- [Background] Crisp M, Starkey KJ, Lane C, Ham J, Ludgate M. Adipogenesis in thyroid eye disease. Invest Ophthalmol Vis Sci. 2000 Oct;41(11):3249-55. PMID 11006210
- [Background] Werner SC. Modification of the classification of the eye changes of Graves' disease. Am J Ophthalmol. 1977 May;83(5):725-7. doi: 10.1016/0002-9394(77)90140-4. PMID 577380
- [Background] Van Dyk HJ. Orbital Graves' disease. A modification of the "NO SPECS" classification. Ophthalmology. 1981 Jun;88(6):479-83. PMID 6894971
- [Background] Gorman CA, Garrity JA, Fatourechi V, Bahn RS, Petersen IA, Stafford SL, Earle JD, Forbes GS, Kline RW, Bergstralh EJ, Offord KP, Rademacher DM, Stanley NM, Bartley GB. A prospective, randomized, double-blind, placebo-controlled study of orbital radiotherapy for Graves' ophthalmopathy. Ophthalmology. 2001 Sep;108(9):1523-34. doi: 10.1016/s0161-6420(01)00632-7. PMID 11535445
- [Background] Bartley GB, Gorman CA. Diagnostic criteria for Graves' ophthalmopathy. Am J Ophthalmol. 1995 Jun;119(6):792-5. doi: 10.1016/s0002-9394(14)72787-4. PMID 7785696
- [Background] Mourits MP, Prummel MF, Wiersinga WM, Koornneef L. Measuring eye movements in Graves ophthalmopathy. Ophthalmology. 1994 Aug;101(8):1341-6. doi: 10.1016/s0161-6420(94)31164-x. PMID 8058278
- [Background] Nugent RA, Belkin RI, Neigel JM, Rootman J, Robertson WD, Spinelli J, Graeb DA. Graves orbitopathy: correlation of CT and clinical findings. Radiology. 1990 Dec;177(3):675-82. doi: 10.1148/radiology.177.3.2243967.
- [Background] Kao SC, Kendler DL, Nugent RA, Adler JS, Rootman J. Radiotherapy in the management of thyroid orbitopathy. Computed tomography and clinical outcomes. Arch Ophthalmol. 1993 Jun;111(6):819-23. doi: 10.1001/archopht.1993.01090060107032. PMID 8512483
- [Background] Prummel MF, Gerding MN, Zonneveld FW, Wiersinga WM. The usefulness of quantitative orbital magnetic resonance imaging in Graves' ophthalmopathy. Clin Endocrinol (Oxf). 2001 Feb;54(2):205-9. doi: 10.1046/j.1365-2265.2001.01220.x. PMID 11207635
- [Derived] Shen S, Fong KS, Wong HB, Looi A, Chan LL, Rootman J, Seah LL. Normative measurements of the Chinese extraocular musculature by high-field magnetic resonance imaging. Invest Ophthalmol Vis Sci. 2010 Feb;51(2):631-6. doi: 10.1167/iovs.09-3614. Epub 2009 Jul 30. PMID 19643971